CLINICAL TRIAL: NCT01686308
Title: The Effect of Cataract on Photoentrainment of the Circadian Rhythm in Humans
Acronym: CIRCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Adam Elias Brøndsted, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRCAT
Record Dates: First submitted 2011-11-30; First posted 2012-09-18 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Cataract
Keywords: cataract; circadian rhythm; pupillometry; blue light transmission; questionnaire; sleep
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Intra Ocular Lens (IOL) (Active Comparator): Standard minimal incision cataract surgery by phacoemulsification and posterior intraocular lens implantation.
  Interventions: Procedure: Conventional Intra Ocular Lens (IOL)
- Yellow Intra Ocular Lens (IOL) (Experimental): Standard minimal incision cataract surgery by phacoemulsification and posterior intraocular lens implantation.
  Interventions: Procedure: Yellow Intra Ocular Lens (IOL)

INTERVENTIONS:
Procedure: Yellow Intra Ocular Lens (IOL) — Standard operation with blue light filter Yellow IOL implantation
  Arms: Yellow Intra Ocular Lens (IOL)
Procedure: Conventional Intra Ocular Lens (IOL) — Standard operation with conventional IOL implantation
  Arms: Conventional Intra Ocular Lens (IOL)

SUMMARY:
Cataract is globally the most common cause of blindness and in Denmark the operation with - 50.000 treatments per year - is the most common eye operation. The cause of cataract is growth and denaturation of the lens proteins. This leads to an increased absorption of blue light and increased light scatter. This may affect newly discovered cells in the retina that are involved in the regulation of the circadian rhythm. When the internal circadian rhythm is not synchronized with the external day and night a phase-shift occurs. Most people know of this discomfort as jet-lag, but the consequences may be much more severe such as heighten risk of cancer and cardiovascular disease.

The goal of this project is to study how the circadian regulating cells of the retina is affected by cataract and by the operation. Cataract patients are studied before and after the operation with questionnaires, hormone and activity measurements and with a specialized pupil measurement that measures the indirect response of the circadian regulating cells to blue light.

Results from this study aim to shed light on the regulatory mechanisms of the eye on the circadian rhythm and how these are affected by cataract. Furthermore, choice of intraocular lens is evaluated. This may have impact on clinical practise especially with regard to choice of intraocular lens and widened indications for cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age related/senile bilateral cataract
* Eligible for phaco-emulsification on both eyes

Exclusion Criteria:

* Known eye disease other than cataract.
* Known systemic disease, which may affect the retina (untreated hypertension, DM etc.)
* Known systemic disease, which may affect the lens.
* Known psychiatric disease.
* Known sleep or circadian rhythm disorder, not caused by lowered blue light transmission by the lens.
* Per- and post operative complications
* Use of drugs that may affect the sleep.

For a subpopulation also:

* Poor cooperation.
* Severe refraction abnormalities.
* Previous eye surgery
* Nystagmus
* Congenital or acquired abnormalities of: eye lids and eye area, cornea or iris.
* Use of medicine that may affect the pupillary response.
* Use of drugs that may affect the pupillary response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pupillary response to blue light | 1 year/1month
  Measurement of the consensual light response to red (630 nm) and blue (470 nm)

SECONDARY OUTCOMES:
Questionnaire | 1year/1month
  Pittsburgh Sleep Quality Index and the Morningness Eveningness Questionnaire
Questionnaire | 1 year/1 month
  Morningness-eveningness questionnaire
Melatonin day variety analysis | 1year/1month
  Salivary samples collected with 4 hour interval during 24 hours. Analyzed for melatonin concentration with Radio Immuno Assay (RIA).
Actigraphy | 1year/1month
  Activity measured during 7 days and 7 nights with the Spectrum Actiwatch, Respironics, Philips

CONTACTS AND LOCATIONS:
Overall Officials: Adam E Brøndsted, MD, Principal Investigator — Glostrup UH
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Denmark